CLINICAL TRIAL: NCT00715702
Title: An Open-Label, Single-Centre, Parallel Group, Phase I Study To Compare the Pharmacokinetics of AZD5672 Single Dose in Patients With Renal Impairment and Healthy Volunteers
Brief Title: Safety Study of AZD5672 in Renally Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Layton, MD, PhD, Medical Science Director, AstraZeneca R&D Alderely Park
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1710C00020; EudraCt nr 2007-007541-
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Renal Impairment
Keywords: AZD5672
MeSH Terms: conditions — Renal Insufficiency | interventions — N-(1-(3-(3,5-difluorophenyl)-3-(4-methanesulfonylphenyl)propyl)piperidin-4-yl)-N-ethyl-2-(4-methanesulfonylphenyl)acetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients with Moderate renal impairment and matched volunteers
  Interventions: Drug: AZD5672
- 2 (Experimental): Patients with Mild or Severe renal impairment and matched volunteers. Type of patient group determined after safety review of 1st group data
  Interventions: Drug: AZD5672

INTERVENTIONS:
Drug: AZD5672 — 100 mg oral single dose

SUMMARY:
The purpose of the study is to investigate the pharmacokinetics of a single dose of AZD5672 in patients with renal impairment by comparing with healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent.
* Females should not be of childbearing potential
* Subjects classified as renally impaired should have been stable (in the Investigator's opinion) for at least 3 months prior to Visit 1.

Exclusion Criteria:

* Patients taking prescription of medications: Pgp substrates, inhibitors and /or inducers, medications that affect creatinine clearance(within 7 days of dosing), atorvastatin >20mg once daily, medications that prolong QT/QTc interval
* Change in dose regimen of prescribed medication and NSAIDs within the 2 weeks before enrolment (renal patients only)
* Participation in another clinical study involving administration of an investigational product in the 3 months prior to treatment (or within 5 half-lives of the last dose of the investigational product, whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during study period

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Rod Hepburn, Study Director — AstraZeneca R&D, Charnwood, UK; Angelika Weil, Principal Investigator — APEX GmbH
Locations (1):
- Research Site, München, Germany